CLINICAL TRIAL: NCT03318627
Title: Influence of Intraoperative Repair Tension on Postoperative Healing of Full-thickness Rotator Cuff Tears
Acronym: TENS-RCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No capacity to conduct the study
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-00236
Record Dates: First submitted 2017-06-29; First posted 2017-10-24 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tension Measuring (Other): Measuring intraoperative tension of rotator cuff tendon with sterile spring Balance.
  Interventions: Device: Sterile Spring Scale

INTERVENTIONS:
Device: Sterile Spring Scale — Measuring intraoperative tension of tendon of rotator cuff tear

SUMMARY:
Relevant problems of rotator cuff repair:

* High retear rate after rotator cuff repair of 13%, despite regard of the criteria for "reparability" of a tear.
* Long and exhausting rehabilitation after rotator cuff repair with an abduction splint for six weeks.

Hypothesis:

The investigators believe that high tension repair has a higher retear rate than low tension repair, regardless of the tear size. The investigators also believe that abduction of the arm can reduce relevant tension on the repair. But not each repair benefits equally from this.

Relevance of this hypothesis:

The ingenious advantage of this new parameter (intraoperative repair tension) is, that it can be influenced. In future, if this hypothesis would be true, the repair tension could be reduced intraoperative by release, side-to-side (margin convergence) repair or medialization of the footprint and thereby convert a high risk to a low risk tension repair.

Moreover, it could be that patients with a low tension repair does not necessarily have to wear an abduction splint. And on the other hand, high tension repair patients should probably wear the abduction splint longer with gradually reduction.

Approach:

The present research plan focused on a new intraoperative (arthroscopic) determinable parameter ("repair tension" on footprint in 0° and 40° abduction) to determine the risk of recurrence after tendon repair in rotator cuff tears, which are pre- and intraoperative defined as "reparable". Therefore, the tension of the repaired tendon is measured intraoperative with a spring balance (newtonmeter) and correlated with the postoperative retear-rate.

• Measure intraoperative repair tension with the arm in 0° and 40° of abduction

DETAILED DESCRIPTION:
How the investigators plan the study:

This is a prospective clinical study, risk category A. It is one-armed (all participants have the same procedure/rehabilitation) and single-blinded (participants doesn't knows the repair tension).

The investigators are an orthopaedic clinic in Zurich (Universitätsklinik Balgrist, Zürich) with about 250 arthroscopic rotator cuff repairs per year. Our plan is to recruit at least 100 participants in a year for this prospective clinical study. The participants have to fulfill the inclusion criterions. The diagnosis for the rotator cuff tears are made on the basis of arthro-MRI scans. The investigators do the operations in our clinic. The entire follow-up is one year for each participant. We plan three regular postoperative consultations. The tendon healing is controlled postoperative by ultrasound (six weeks and 4 month postoperative) and by MRI (one year postoperative).

Visit 0: participant recruitment:

The participants who are suitable for the study, will be recruited in the clinic for the study. They are aware of the essential information and the process and have 14 days time to read the information paper.

Visit 1: preoperative phase:

The following parameters are collected by default:

* Constant score
* Begin of symptoms (subjective shoulder value, visual analogue scale)
* Questionnaire
* Arthro-MRI (fatty infiltration, tear size, tendon retraction, length of central tendon)
* RX (Critical Shoulder Angle)

Visit 2: intraoperative phase:

The intraoperative procedure is standardized:

Postoperative immobilisation in an abduction splint in 40° abduction with passive mobilisation (physiotherapy) without adduction for six weeks.

Visit 3: 6 weeks postoperative phase:

The following parameters are collected by default:

* Clinical examination
* Subjective shoulder value
* Pain-VAS
* Questionnaire
* Complications
* Ultrasound (retear yes/no) The abduction splint is removed. Other six weeks mobilisation active and active-assisted without weights and strength until the 12th week (clinic standard).

Visit 4: 4 months postoperative phase:

The following parameters are collected by default:

* Clinical examination
* Active ROM (abduction, flexion, external rotation)
* Passive ROM (glenohumeral abduction, external rotation)
* Subjective shoulder value
* Pain-VAS
* Questionnaire
* Complications
* Ultrasound (retear yes/no) There is an increase in strength and agility

Visit 5: 1 year postoperative phase:

The following parameters are collected by default:

* Clinical examination
* Passive ROM (glenohumeral abduction, external rotation)
* Subjective shoulder value
* Pain-VAS
* Constant score
* Questionnaire
* Complications
* MRI (fatty infiltration)
* X-ray (critical shoulder value) The study is finished for the patient

How the investigators can realise the aims:

Aim 1: Correlation of intraoperative repair tension in 0° and 40° abduction on footprint with postoperative healing.

The investigators measure intraoperative repair tension for each participant in 0° and 40° abduction in gram with a spring balance. Then, measurement of healing rate of these tendon reconstructions over one year. The investigators do three regular follow-ups. In week 6 and month 4, control of healing with ultrasound and one year postoperative with an MRI scan. Intraoperative repair tension is correlated with retear rate. Cut-off value to separate high risk and low risk tension repairs is evaluated.

Aim 2: Correlation of other parameters with postoperative healing: The investigator correlate other parameters with the postoperative healing. Following parameters are collected in preoperative MRI scans: tear size in cm, tear retraction in cm, central tendon length in cm, fatty infiltration with the classification of Goutallier I-IV. In preoperative x-rays we measure the critical shoulder angle in degree. Intraoperative measurement of: tendon quality in four stages and the tear pattern visual (see above, "Visit 2").

Aim 3: Can intraoperative repair tension be predicted preoperative by MRI findings?: For this question, measurement of following parameters: tendon size in cm, tendon retraction in cm, length of central tendon in cm and fatty infiltration with the classification of Goutallier I-IV. Statistical evaluation with correlation of intraoperative repair tension with these MRI findings.

Aim 4: Correlation of high repair tension with pain: Correlation of pain with repair tension. Measurement of pain in each consultation with a visual analogue scale from 0-10 (0 no pain, 10 very much pain). Measurement range of motion of the participants (active and passive) and correlate stiffness with pain and with repair tension.

Aim 5: Correlation of repair tension with postoperative muscle atrophy, fatty infiltration and tendon length: Measurement of muscle atrophy, fatty infiltration and tendon length in the MRI scan preoperative and one year postoperative to compare. The muscle atrophy is quantified with tangent sign and occupation ratio. Fatty infiltration with the classification of Goutallier and tendon length in cm. Then, correlation pre- and postoperative changes with the repair tension.

Aim 6: Lower retear rate in type B- and C-reconstruction compared to type A- reconstruction? (type A-C) If possible, the investigators want to correlate different reconstruction types (A-C) with similar tension repairs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male/female from 18-99 years
* All arthroscopic reparable transmural supra-/infraspinatus tears
* German speaking

Exclusion Criteria:

* Previous operation on the ipsilateral rotator cuff
* Irreparable rotator cuff tear (supra- and / or infraspinatus and / or subscapularis)
* static antero-superior subluxation of humeral head
* dynamic antero-superior subluxation of humeral head
* pseudoparalysis for anteflexion, hornblow sign, dropping- arm sign
* fatty infiltration goutallier 3-4 (MRI)
* reduced acromiohumeral distance <7mm (RX)
* intraoperative not reparable
* Mild/severe osteoarthritis (RX, Hamada II-IV)
* Inability of patient (language problems, mental illness, dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Tendon tension | during surgery
  Measuring tendon Tension according to the footprint in 0° and 45° abduction with a Newtonmeter.

SECONDARY OUTCOMES:
Rotator cuff re-tear | one year
  Evaluation re-tear of repaired rotator cuff in MRI scan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le BT, Wu XL, Lam PH, Murrell GA. Factors predicting rotator cuff retears: an analysis of 1000 consecutive rotator cuff repairs. Am J Sports Med. 2014 May;42(5):1134-42. doi: 10.1177/0363546514525336. Epub 2014 Apr 18. PMID 24748610
- [Background] Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40. doi: 10.2106/JBJS.D.02035. PMID 15930531
- [Background] Thomazeau H, Boukobza E, Morcet N, Chaperon J, Langlais F. Prediction of rotator cuff repair results by magnetic resonance imaging. Clin Orthop Relat Res. 1997 Nov;(344):275-83. PMID 9372778
- [Background] Meyer DC, Wieser K, Farshad M, Gerber C. Retraction of supraspinatus muscle and tendon as predictors of success of rotator cuff repair. Am J Sports Med. 2012 Oct;40(10):2242-7. doi: 10.1177/0363546512457587. Epub 2012 Aug 27. PMID 22926748
- [Background] Liem D, Lichtenberg S, Magosch P, Habermeyer P. Magnetic resonance imaging of arthroscopic supraspinatus tendon repair. J Bone Joint Surg Am. 2007 Aug;89(8):1770-6. doi: 10.2106/JBJS.F.00749. PMID 17671017